CLINICAL TRIAL: NCT03557554
Title: A Prospective Feasibility Study Investigating Primary Preventive Ability of Massage Therapy of Paclitaxel-Induced Peripheral Neuropathy in Patients With Newly Diagnosed Breast Cancer Scheduled to Undergo a Paclitaxel Based Regimen
Brief Title: Investigating the Preventative Ability of Massage Therapy on Paclitaxel Induced Peripheral Neuropathy
Acronym: PIPN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: feasability and recruitment issues
Sponsor: Bryan Schneider (Other)
Collaborators: Massage Therapy Foundation (Other)
Responsible Party: Sponsor-Investigator, Bryan Schneider, Principal Investigator, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IUSCC-0616 (1709077419)
Record Dates: First submitted 2018-04-11; First posted 2018-06-15 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Neuropathy; Neuropathy;Peripheral
Keywords: Massage; Breast Cancer; Neuropathy
MeSH Terms: conditions — Breast Neoplasms; Neuritis | interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Massage Therapy (Experimental): Subjects who are planning treatment with paclitaxel as part of their standard of care treatment will receive a 20 minute massage prior to each paclitaxel infusion.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — A 20 minute massage protocol will be administered in a chair by a licensed massage therapist no more than 24 hours prior to each paclitaxel infusion.

SUMMARY:
Feasibility study to examine the preventative ability of massage therapy on paclitaxel induced peripheral neuropathy in breast cancer

ELIGIBILITY:
Inclusion Criteria:

1) Breast cancer diagnosis 2) Planning to receive chemotherapy treatment with paclitaxel in the curative setting (adjuvant or neoadjuvant) on a weekly or bi-weekly schedule

Exclusion Criteria:

1)Diabetes or other neurological disorder 2) Current or previous peripheral neuropathy 3)Previous treatment with paclitaxel 4)Active deep vein thrombosis (DVT) within last 12 months or history of untreated lower extremity DVT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of Recruitment | 1 year
  rate of enrollment
Feasibility of Retention | 1 year
  rate of drop out or consent withdraw

SECONDARY OUTCOMES:
Incidence of paclitaxel induced peripheral neuropathy | 10 months
  incidence of paclitaxel induced peripheral neuropathy as measured using the Assessment of Cancer Therapy-Neurotoxicity (FACT-Ntx) questionaire
Severity of paclitaxel induced peripheral neuropathy | 10 months
  severity of paclitaxel induced peripheral neuropathy measured by Assessment of Cancer Therapy-Neurotoxicity (FACT-Ntx) questionnaire
Rate of pharmacological interventions | 10 months
  pharmacological interventions for paclitaxel induced peripheral neuropathy
Paclitaxel dose modification | 4 months
  rate of dose modifications to paclitaxel treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Schneider, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No